CLINICAL TRIAL: NCT03312504
Title: Evaluating the Effectiveness of Neuromuscular Training in Decreasing the Risk of Sport and Recreational Injuries and Improving Healthy Outcomes in Junior High School Students
Brief Title: Implementing a School Prevention Program to Reduce Injuries Through Neuromuscular Training
Acronym: iSPRINT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Calgary Board of Education (Other); Calgary Catholic School District (Other); Ever Active Schools (Unknown); Policywise for Children and Families (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB14-0470
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Wounds and Injuries; Adolescent; Athletic Injuries; Sport Injury; Sports Injuries in Children
Keywords: sport injury; injury prevention; fitness; neuromuscular training; implementation
MeSH Terms: conditions — Wounds and Injuries; Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Upon enrolment into the study, a school will be randomly assigned to the intervention (neuromuscular training warm-up) or control group (standard-of-practice warm-up). Schools that have been randomized to the control arm will be invited to participate in the study in the following year as an intervention school. Schools that have been randomized to the intervention arm will be invited to participate in the study in the following year as a maintenance school (will continue with the intervention).
Who Masked: Participant, Investigator
Masking Description: Participants (teachers and students) are not aware of what arm they are randomized to; however, they are aware that there are two arms. The primary investigators performing the analysis and overseeing all decisions are blinded to the schools receiving the intervention vs control program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Training Warm-up (Experimental): Schools randomized to the intervention arm receive a workshop outlining a neuromuscular training program to be used as a warm-up for 15 minutes at the beginning of each physical education class. The warm-up consist of high-intensity aerobic, strengthening, agility, plyometric, and balance components. The workshop is designed to last two hours, and includes a video outlining the warm-up components, practice time, and group discussions for action planning to address potential barriers to the program.
  Interventions: Other: Neuromuscular training program
- Control Standard-of-practice Warm-up (Placebo Comparator): Schools randomized to the control arm receive a workshop outlining a standard-of-practice program to be used as a warm-up for 15 minutes at the beginning of each physical education class. The warm-up consists of aerobic exercises and static stretching. The workshop is designed to last one hour, and includes an explanation and demonstration of the exercises, but no video or practice time.
  Interventions: Other: Standard-of-practice Warm-up (Control)

INTERVENTIONS:
Other: Neuromuscular training program — This is a 15-minute warm-up program designed to be implemented at the beginning of junior high school physical education classes. This warm-up is comprised of 15 components; nine of which are aerobic exercises (forward running, forward run with skipping, forward run with knee lifts, forward run with heel kicks, sideways shuffles, zigzag running, forward running with intermittent stops, speed runs, and squat/skate jumps), and six of which are balance/strengthening exercises (front plank, side plank, nordic hamstring exercise, lunges, balancing on the wobble board, and balancing on foam balance pads).
  Arms: Neuromuscular Training Warm-up
Other: Standard-of-practice Warm-up (Control) — This is a 15-minute warm-up program designed to be implemented at the beginning of junior high school physical education classes. This warm-up is comprised of 16 components; seven of which are aerobic exercises (forward running, forward running with arm swings, side shuffling, lunging, skipping, arm running with arm swings, and cool-down running), and nine of which are static stretching exercises (standing quadriceps, standing hamstrings, standing calf, standing groin, rotating ankle, lunges, standing shoulder, standing triceps, standing neck).
  Arms: Control Standard-of-practice Warm-up

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a neuromuscular training program in decreasing sport and recreational injuries and improving healthy outcomes in junior high school students (grades 7 to 9). The neuromuscular training program is implemented as a 15-minute warm-up at the beginning of the students' physical education classes over a three-month period. This study is a randomized controlled trial design, involving twelve schools over a three-year period. Upon enrolment into the study, schools are randomly assigned to the intervention (neuromuscular training) group, or the control group. The control group includes a standard-of practice warm-up consisting of aerobic components and static stretching.

A study athletic therapist visits the schools each week to assess and record information on any injuries sustained by study participants. Baseline health and physical fitness is measured at baseline, and again at 3-month follow-up in study participants to assess changes over the course of the program.

ELIGIBILITY:
Inclusion Criteria:

SCHOOLS

* junior high schools with a minimum of two physical education classes per week, per class
* physical education classes that are taught or co-taught by a physical education specialist

SUBJECTS

* students aged 11-15 who are fully participating in physical education curriculum at baseline
* students who return completed assent and parental consent forms

Exclusion Criteria:

SCHOOLS

* schools that are culturally distinct
* schools that have students that are of single sex
* schools that cater to students with special needs
* schools with incomplete grades

SUBJECTS

* history of musculoskeletal disorders or medical condition that prevents participation in regular physical education curriculum
* history of musculoskeletal injury within 6 weeks prior to study commencement that restricts full participation in physical education
* at least 80% of participation in physical education classes over the course of the study

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1067 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Sport or recreational injury | Injuries are recorded if sustained at any point over the course of the study (each school participates for 3 months).
  Any injury sustained through a sport or recreational activity that resulted in time loss from physical activity participation (unable to return to the same session or missed at least one day of participation), or required medical attention.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) | Changes over a 3-month period.
  Height (cm) and weight (kg) are measured at baseline, and again post-intervention at 3-months. Height and weight are used to calculate body mass index, calculated as: weight(kg)/height(m)^2
Changes in waist circumference | Changes over a 3-month period.
  Waist circumference (cm) is measured at baseline, and again at 3-month follow-up once the intervention in complete. Waist circumference is measured following the Canadian Society for Exercise Physiology-Canadian Physical Activity, Fitness and Lifestyle Approach protocol: circumference is measured at the midpoint between the anterior superior iliac spine and the bottom of the ribs, at the end of a normal expiration while the participant crosses their arms over their chest.
Changes in vertical jump height | Changes over a 3-month period
  Vertical jump height (cm) is measured at baseline, and again post-intervention at 3-month follow-up. The height is calculated as the difference (in cm) between the standing reach height, and the maximum reach measured while jumping from the best of three trials.
Changes in VO2max | Changes over a 3-month period
  The PACER 20-m shuttle run is used to indirectly measure VO2max. Participants run the 20-m shuttle run at baseline, and again post-intervention at 3-month follow-up. Their score (recorded in number of laps) and used in a regression equation to predict maximal oxygen consumption.
Changes in timed unipedal eyes-closed dynamic balance | Changes over a 3-month period
  Balance times are measured at baseline, and again post-intervention at 3-month follow-up. The participant stands on an unstable foam pad (Airex balance pad) on one foot, with their eyes closed and hands on their hips. Time is recorded in seconds for each foot, and the best of three trials on each foot is used to assess changes.
Changes in Y-balance reach distance | Changes over a 3-month period
  Normalized composite reach distance is measured using the Y-balance test at baseline and again post-intervention at 3-month follow-up. The participant balances on one foot while pushing a sliding block as far as they can with their other foot, while maintaining balance. This is repeated for a total of three reach directions on each foot: anterior, postero-lateral, and postern-medial. Reach distances for each of the three directions are normalized as a percentage of leg length of the reaching leg, and summed to produce a normalized composite reach distance.

REFERENCES:
- [Result] Emery CA, van den Berg C, Richmond SA, Palacios-Derflingher L, McKay CD, Doyle-Baker PK, McKinlay M, Toomey CM, Nettel-Aguirre A, Verhagen E, Belton K, Macpherson A, Hagel BE. Implementing a junior high school-based programme to reduce sports injuries through neuromuscular training (iSPRINT): a cluster randomised controlled trial (RCT). Br J Sports Med. 2020 Aug;54(15):913-919. doi: 10.1136/bjsports-2019-101117. Epub 2019 Dec 10. PMID 31822477